CLINICAL TRIAL: NCT05113316
Title: Mental Health Resources for Frontline Healthcare Workers Using the Messy Memories App
Brief Title: Mental Health Resources for Frontline Healthcare Workers
Acronym: Messy-Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sheila Rauch, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003287
Record Dates: First submitted 2021-11-01; First posted 2021-11-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Mental Health
Keywords: Mental Health in Healthcare Workers; Stress-related problems; Frontline Workers
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Complete research clinical trial (RCT) with a sample of frontline healthcare workers to examine the Messy Memories app versus treatment as usual (TAU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Messy Memories App Group (Experimental): Subjects will download and have access to the Messy Memories application in addition to completing self-report measures electronically at pre-determined time points. While the subject uses the app, the participant will input information related to their mood over the past few days (affect rating sliders), their level of distress before and after the memory processing, answers to questions about revisiting the memory, answers to questions in the social connection and self-care modules including assessment of, for example, sleep pattern, eating habits, and exercise habits.
  The Messy Memories app will also collect data on how frequently and for how long each participant uses the app. Each response will trigger a prompt within the app, and will be recorded with a timestamp (date and time) to indicate when the participant provided a particular response. For all participants, self-report measures will be collected at weeks 4, 8, 12, and 16.
  Interventions: Behavioral: Messy Memories App
- Treatment as usual (TAU) Group (No Intervention): Subjects will not receive any study treatments or have access to the app but may seek standard treatment if they choose, in addition to completing self-report measures. For 8 weeks, TAU group will participate in the study under treatment as usual. For weeks 9-16, the TAU group will then switch and have full access to the Messy Memories App to review and use for a limited amount of time. Subjects will download and have access to the Messy Memories application in addition to completing self-report measures electronically at pre-determined time points. While the subject uses the app, the participant will input information related to their mood over the past few days, their level of distress before and after the memory processing, answers to questions about revisiting the memory, answers to questions in the social connection and self-care modules including assessment of, for example, sleep pattern, eating habits, and exercise habits.

INTERVENTIONS:
Behavioral: Messy Memories App — The Messy Memories mobile app is an intervention targeting stress-related problems based on practices with proven effectiveness, to overcome barriers and provide access to evidence-informed intervention strategies aimed to improve mental health in frontline healthcare workers.
  The app allows the user to self-administer exposure therapy techniques outside of the traditional psychotherapy context. The Messy Memories app was initially released in a written form for self-help, but with widespread use of smartphones, a mobile application has the potential to further reduce barriers and increase access to care among frontline healthcare workers. The current study proposes to examine this newly developed application for usability and feasibility in a small sample of frontline healthcare workers (Phase I) and then test efficacy of the application in a larger-scale RCT (Phase II) where the application will be compared to a TAU condition.
  Arms: Messy Memories App Group

SUMMARY:
The proposed study is designed to test and optimize the Messy Memories mobile application as an intervention. The Messy Memories mobile intervention is designed to target stress-related problems based on practices with proven effectiveness. By utilizing a mobile application intervention, this study aims to overcome barriers and provide access to evidence-informed intervention strategies that will likely improve mental health in frontline healthcare workers.

DETAILED DESCRIPTION:
A previous Phase I of this study aimed to test usability (Phase I) of the mobile application. Following this Phase I, this current study Phase II is aimed to test effectiveness of the mobile application ("Messy Memories") in frontline healthcare workers at Emory. Considering current increases in mental health concerns and shortage of mental healthcare providers, the Messy Memories app was designed to target stress-related problems and provide frontline healthcare workers easy access to a mental health intervention that is evidence-informed.

The population to be studied includes adults (ages 18-89 years) employed at Emory Healthcare/University in Atlanta, Georgia. Potentially vulnerable participants that will be enrolled include pregnant women.

Participants will be recruited via email blast and fliers posted in clinics at Emory. These postings will include an electronic link that the potential participant can use to contact the study staff. Informed consent for Phase I will be obtained via online survey, and for Phase II informed consent will be obtained in written form (electronical consent document). This is a minimal risk and contact-less study.

The data collected is not publicly available. Data that is collected as part of this study will be de-identified before use in any analysis or publication. Research study staff will have access to participant names and contact information for the duration of their study participation for compensation purposes. Only members of the research study staff will have access to the code that links identifiers to subjects. Privacy of existing data is not a concern for this study. No HIPAA waiver is needed for this study.

Contact with participants will occur solely electronically via electronic surveys (in REDCap), emails, phone, and focus group (group discussion) via Zoom. Participants will be able to complete study tasks at any remote location that is most convenient for them. Participants will be advised to complete study tasks in the app in a private space. General scope of topics areas includes stress, depression, anxiety, traumatic experiences, burnout, wellbeing, and health behaviors.

Phase I participants will be expected to spend approximately 2 hours on study tasks, not including app use. Time spent on app use (during 2 weeks) will be at the discretion of the participant. Phase II participants will be expected to spend approximately 5 hours on study tasks, also not including app use which will be at the participant's discretion (during 16 weeks).

A participant will be identified throughout the central database by his or her unique subject identification number (SID). All research information will be stored in password-protected folders on secure and HIPAA-compliant servers that can only be accessed by the study staff and non-Emory co-investigators who sign Data Use Agreements.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and female frontline healthcare employees between ages of 18 and 89.
* Participants must be employed at Emory Healthcare/University
* Participants must comprehend his or her role in the study and the risks involved in

Exclusion Criteria:

* Not fluent in English language
* Individuals who identify concerns that indicate high risk for suicide or self-harm behaviors
* Individuals who deny any stressful or traumatic experiences in their lifetime
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Community Participation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Affect Assessments with Messy Memories Apps | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  While the participant uses the Messy Memories app, the participant will input information related to their mood over the past few days (affect rating sliders), their level of distress before and after the memory processing, answers to questions about revisiting the memory

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The PHQ-9 is a nine item self-report of general depression and distress. Scores are assessed by adding the columns and then multiplying the sum of the columns by 1, 2, or 3. Several studies support its validity, feasibility, and its capacity to detect changes of depressive symptoms over time
Change in PTSD Checklist for DSM-5 (PCL-5) | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The PCL-5 is a 20-item self-report measure designed to assess the Diagnostic and Stastistical Manual of Menatl Health's symptoms (DSM-5) of PTSD.
Life Events Checklist (LEC) for DSM-5 | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The LEC is a 17-item self-report measure designed to inventory stressful/traumatic life events
Change in The Alcohol Use Disorders Identification Test: Self-Report Version (AUDIT) | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The AUDIT is a 10-item self-report measure designed to screen for problematic alcohol use (developed by the World Health Organization; WHO)
Change in Maslach-Burnout Inventory | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The Maslach-Burnout Inventory is a 22-item self-report measure designed to inventory burnout within the work environment as defined by the WHO.
Change in Perceived Stress Scale (PSS): | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The PSS is a 10-item self-report measure designed to examine frequency of thoughts and feelings related to perceived stress. The measure has been validated and widely used in the general population.
Change in The Connor-Davidson Resilience Scale Brief Version (CD-RISC 10) | At baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  The CD-RISC 10 is a 10-item measure of resilience following stressful experiences
How frequently is the app used | From baseline to week 16
  each response to a prompt within the app will be recorded with a timestamp (date and time) to indicate when the participant provided a particular response.
For how long is the app used | From baseline to week 16
  each response to a prompt within the app will be recorded with a timestamp (date and time) to indicate when the participant provided a particular response.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila A.M. Rauch, PhD, Principal Investigator — Emory University
Locations (1):
- 12 Executive Park, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The results of the study will not be shared with participants at the individual level. Once the aggregate data are analyzed, participants may request the study results from the research team. A member of the research team will make these results available after the completion of the study.